CLINICAL TRIAL: NCT00136201
Title: A Multicenter, Randomized, Open-Label Comparison of the Safety and Efficacy of Tigecycline> vs Imipenem/Cilastatin to Treat Complicated Intra-Abdominal Infections in Hospitalized Chinese Subjects
Brief Title: Study Comparing Tigecycline and Imipenem/Cilastatin in Chinese Subjects With Complicated Intra-Abdominal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-316
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Abdominal Abscess
Keywords: Peritonitis; Community-Acquired Infections; Cross Infection
MeSH Terms: conditions — Abdominal Abscess; Peritonitis; Community-Acquired Infections; Cross Infection | interventions — Tigecycline

ARMS (1):
- 1 (Experimental): armDesc1
  Interventions: Drug: tigecycline

INTERVENTIONS:
Drug: tigecycline

SUMMARY:
The primary objective of this study is to compare the safety and efficacy of an experimental antibiotic to a marketed antibiotic in the treatment of Chinese subjects with complicated intra-abdominal infections. <br />

ELIGIBILITY:
Inclusion Criteria:

· Hospitalized male or female subjects over 18 years of age

Exclusion Criteria:

· Subjects with any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy or follow-up visits could be completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Clinical response for all microbiologically evaluable and microbiologically modified intent-to-treat subjects at the test-of-cure visit

SECONDARY OUTCOMES:
Microbiological response at the subject and pathogen level and evaluation of microbiological data, such as decreased susceptibility, response rates by baseline isolate and minimal inhibitory concentration (MIC) values and susceptibility data by isolate

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com
Locations (6):
- China (6):
  - Guoxuexiang, Chengdu
  - Shengyang, Liaoning
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
  - Wuhan

REFERENCES:
- [Derived] Chen Z, Wu J, Zhang Y, Wei J, Leng X, Bi J, Li R, Yan L, Quan Z, Chen X, Yu Y, Wu Z, Liu D, Ma X, Maroko R, Cooper A. Efficacy and safety of tigecycline monotherapy vs. imipenem/cilastatin in Chinese patients with complicated intra-abdominal infections: a randomized controlled trial. BMC Infect Dis. 2010 Jul 21;10:217. doi: 10.1186/1471-2334-10-217. PMID 20663130
- [Derived] Fomin P, Koalov S, Cooper A, Babinchak T, Dartois N, De Vane N, Castaing N, Tellado J; 301 And 306 Study Groups. The efficacy and safety of tigecycline for the treatment of complicated intra-abdominal infections - the European experience. J Chemother. 2008 Oct;20 Suppl 1:12-9. doi: 10.1179/joc.2008.20.Supplement-1.12. PMID 19036670